CLINICAL TRIAL: NCT00012129
Title: Phase I/II Clinical and Pharmacological Study of Liposomal Annamycin in Anthracycline-Resistant Breast Cancer
Brief Title: Chemotherapy in Treating Patients With Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068486; NYU-9851; NCI-G01-1914
Record Dates: First submitted 2001-03-03; First posted 2004-04-20 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male

INTERVENTIONS:
Drug: liposomal annamycin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of annamycin liposomal in treating patients who have locally advanced or metastatic breast cancer that has not responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the observed anti-tumor activity of annamycin liposomal in patients with anthracycline-resistant locally advanced or metastatic breast cancer. II. Determine the qualitative and quantitative toxicity and reversibility of toxicity of this regimen in these patients. III. Determine the clinical pharmacology of this regimen in these patients. IV. Determine the rationale for the dose and chosen schedule of this regimen in these patients.

OUTLINE: Patients receive annamycin liposomal IV over 60 minutes on day 1. Treatment continues every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 14-30 patients will be accrued for this study within 7-30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of locally advanced or metastatic breast cancer High likelihood of anthracycline resistance due to prior anthracycline exposure in the adjuvant or metastatic setting Prior anthraquinone (e.g., mitoxantrone) insufficient Prior cumulative anthracycline dose limited to doxorubicin-equivalent 350 mg/m2 by IV bolus or 450 mg/m2 by prolonged (at least 48 hours) infusion Measurable or evaluable disease Brain metastases treated by prior surgery and/or radiotherapy allowed if neurologic status stable 2 weeks after discontinuation of dexamethasone Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Male or female Menopausal status: Not specified Performance status: Zubrod 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute granulocyte count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No history of heart failure Ejection fraction at least 55% by 2-dimensional echocardiogram Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception Other prior malignancy allowed if curatively treated and there is clear diagnosis of metastatic breast cancer requiring treatment

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent prophylactic filgrastim (G-CSF) Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosourea) and recovered Endocrine therapy: See Disease Characteristics Radiotherapy: See Disease Characteristics At least 3 weeks since prior radiotherapy and recovered Surgery: See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-09; Primary Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D. Volm, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States